CLINICAL TRIAL: NCT03595228
Title: A Phase 2 Trial of BN-Brachyury and Radiation Therapy in Patients With Advanced Chordoma
Brief Title: BN Brachyury and Radiation in Chordoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRACHY-CHOR-001
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Chordoma
MeSH Terms: conditions — Chordoma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BN-Brachyury plus radiation (Experimental): BN-Brachyury as both MVA and FPV are given before radiation, and followed by FPV-Brachyury
  Interventions: Biological: BN-Brachyury plus radiation

INTERVENTIONS:
Biological: BN-Brachyury plus radiation — MVA-BN-Brachyury injections will be given on day 0 and 14. FPV-Brachyury injection will be given on day 28, followed by radiation on days 42 through approximately day 70. FPV-Brachyury will then be given two weeks after radiation then every 6-12 weeks through 110 weeks after radiation is complete.

SUMMARY:
The goal of this study is to determine if the combination of BN-Brachyury plus radiation therapy can induce objective radiographic response rate (ORR) in patients, using a Simon 2-stage optimal design. In stage 1, a minimum of threshold of activity is needed to proceed to stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed chordoma
* Patients must have measurable disease by RECIST 1.1
* Patients must be scheduled to have radiation therapy to at least 1 target lesion.
* Age ≥12 years
* Patients must have normal organ and marrow function
* Must have recovered completely from any reversible toxicity associated with recent therapy.
* There should be a minimum of 2 weeks from any chemotherapy, small molecule/targeted therapy, immunotherapy and/or radiation prior to enrolment
* Females of childbearing potential and male partners of Females of childbearing potential must agree to use effective birth control or abstinence from screening to after the last vaccination therapy

Exclusion Criteria:

* Concurrent treatment for cancer, with specific exceptions noted in the inclusion criteria
* Chronic hepatitis B or C infection.
* Any significant disease, that in the opinion of the investigator may impair the patient's tolerance of trial treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding, or rendering of informed consent.
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity.
* Concurrent use of systemic steroids, except for physiological doses of systemic steroid replacement or local steroid use.
* Patients who are receiving any other investigational agents within 28 days before start of trial treatment.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to MVA-BN/FPV-Brachyury or other agents used in trial. History of allergic reactions to aminoglycoside antibiotic or egg products.
* Serious or uncontrolled intercurrent illness, included but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with trial requirements.
* Pregnant women are excluded from this trial due to the unknown effects of the BN-Brachyury on the fetus or infant.
* HIV-positive patients are ineligible because of the potential for decreased immune response to the vaccine.
* Significant cardiovascular disease, which includes but is not limited to New York Heart Association Heart Failure Class II or greater, myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cote, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Mayo Clinic, Arizona, Phoenix, Arizona
  - Mayo Clinic, Florida, Jacksonville, Florida
  - Massachusetts General Hospital, Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BN-Brachyury Plus Radiation
Started | 29
Completed | 10
Not Completed | 19
Not completed — Death | 2
Not completed — Lack of Efficacy | 13
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set consists of all subjects who have enrolled and received any dose of MVA-BN Brachyury or FPV-Brachyury
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29
HIV Antibody [Count of Participants; unit: Participants]
  Positive | 0
  Negative | 29
Hepatitis B Surface [Count of Participants; unit: Participants]
  Positive | 0
  Negative | 29
Hepatitis C Virus [Count of Participants; unit: Participants]
  Positive | 0
  Negative | 29
ECOG Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status. Grade 0 = Fully active, able to carry on all pre-disease performance without restriction. Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. Grade 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 12
    1 | 17
    2 | 0
Historical Classification [Count of Participants; unit: Participants]
  Classical | 26
  Chondroid | 0
  Not Reported | 3
Primary Tumor Site [Count of Participants; unit: Participants]
  Clival | 3
  Mobile Spine | 8
  Sacral | 18
Disease Status at Diagnosis [Count of Participants; unit: Participants]
  Localized | 20
  Locally Advanced | 7
  Metastatic | 2
Current Disease Status [Count of Participants; unit: Participants]
  Localized | 0
  Locally Advanced | 5
  Metastatic | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Rate of subjects achieving a best response of either Complete Response or Partial Response per modified RECIST v1.1. A modified RECIST v1.1 assessment is based on targeted radiated lesion(s). Progression of a non-target lesion does not result in disease progression by the modified RECIST evaluation for this trial. Assessment for targeted radiated lesion(s): Complete Response (CR)=Disappearance of all target radiated lesions; Partial Response (PR)= >=30% decrease in the sum of the longest diameter of target radiated lesions; Progressive Disease (PD) = >=20% increase in the sum of the longest diameter of target radiated lesions, Stable Disease (SD)=-30%<sum of the longest diameter of target radiated lesions<20%.
Time Frame: Within 12 months post-completion of radiation on target lesion(s) based on modified RECIST v1.1
Population: Evaluable Analysis Set conisits of subjects who have completed two prime doses of MVA-BN-Brachyury and one booster dose of FPV-Brachyury prior to radiation, have completed radiation therapy, have at least 3 out of 4 booster doses of FPV-Brachyury in 14 weeks after radation, have both baseline and at least one post-baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan for objective tumor evaluation.
Measure: Number (90% Confidence Interval); unit: percentage of subjects with OR
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 26
percentage of subjects with OR | 7.7 [2.6 to 20.8]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Kaplan-Meier of the time interval from first treatment to objective tumor progression based on modified RECIST v1.1 or death. A modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) based on targeted radiated lesion(s) will be used. Progression will be defined as a 20% increase in the sum of the longest diameter of target radiated lesions in this trial, and a progression of a non-target lesion does not result in disease progression by the modified RECIST evaluation used for this trial.
Time Frame: Time from the day of first treatment to the start of disease progression or death, whichever occurs first up to 30 days after last tumor assessment visit. Data were collected up to 29 months.
Population: Evaluable Analysis Set consists of subjects who have completed two prime doses of MVA-BN-Brachyury and one booster dose of FPV-Brachyury prior to radiation, have completed radiation therapy, have at least 3 out of 4 booster doses of FPV-Brachyury in 14 weeks after radation, have both baseline and at least one post-baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan for objective tumor evaluation.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 26
Weeks | NA [51.29 to NA] — It is NA because there are insufficient number of participants with events and hence median and upper 95% confidence interval are not evaluable.

3. Secondary Outcome: Baseline and Overall Treatment Period Change From Baseline Brief Pain Improvement-Short Form Best Observed Scores
Description: Pain intensity and pain interference scores are summarized. Pain intensity scores includes pain items "Worst Pain in the Last Week", "Least Pain in the Last Week", and "Average Pain in the Last Week" and "Pain Right Now". Composite pain severity score (a mean severity score of the four pain items listed before). Composite pain interference score (a mean of the seven interference items). This will be calculated if at least four of the seven interference items have been completed on a given administration. Pain scores range from 0 to 10 with a score of 10 is the worst pain imaginable and a score of 0 is no pain. Best observed scores is the lowest score value observed.
Time Frame: Overall Treatment Period: The time from the day of first treatment to the last scheduled trial visit, approximately 30 days after the last treatment visit. Data were collected up to 29 months.
Population: Evaluable Analysis Set consists of subjects who have completed two prime doses of MVA-BN-Brachyury and one booster dose of FPV-Brachyury prior to radiation, have completed radiation therapy, have at least 3 out of 4 booster doses of FPV-Brachyury in 14 weeks after radiation, have both baseline and at least one post-baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan for objective tumor evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 26
score on a scale
  Worst Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Worst Pain in the Last Week - Baseline | 4 (3.46)
  Least Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Least Pain in the Last Week - Baseline | 1.5 (1.81)
  Average Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Average Pain in the Last Week - Baseline | 2.4 (2.13)
  Pain Right Now - Baseline: number analyzed (Participants) | 21
  Pain Right Now - Baseline | 2 (1.99)
  Composite Pain Severity Score - Baseline: number analyzed (Participants) | 21
  Composite Pain Severity Score - Baseline | 2.476 (2.1779)
  Composite Pain Interference Score - Baseline: number analyzed (Participants) | 21
  Composite Pain Interference Score - Baseline | 2.869 (2.7136)
  Worst Pain in the Last Week - Overall Treatment Period | 2.3 (1.0)
  Least Pain in the Last Week - Overall Treatment Period | 0.8 (0.91)
  Average Pain in the Last Week - Overall Treatment Period | 1.5 (1.53)
  Pain Right Now - Overall Treatment Period | 1.2 (1.43)
  Composite Pain Severity Score - Overall Treatment Period | 1.625 (1.6737)
  Composite Pain Interference Score - Overall Treatment Period | 1.451 (2.0962)
  Worst Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Worst Pain in the Last Week - Change from Baseline in Overall Treatment Period | -1.4 (1.75)
  Least Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Least Pain in the Last Week - Change from Baseline in Overall Treatment Period | -0.7 (1.35)
  Average Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Average Pain in the Last Week - Change from Baseline in Overall Treatment Period | -0.8 (1.03)
  Pain Right Now - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Pain Right Now - Change from Baseline in Overall Treatment Period | -0.8 (0.81)
  Composite Pain Severity Score - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Composite Pain Severity Score - Change from Baseline in Overall Treatment Period | -0.75 (1.0577)
  Composite Pain Interference Score - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Composite Pain Interference Score - Change from Baseline in Overall Treatment Period | -1.127 (1.4096)

4. Secondary Outcome: Baseline and Overall Treatment Period Change From Baseline Brief Pain Improvement-Short Form Worst Observed Scores
Description: Pain intensity and pain interference scores are summarized. Pain intensity scores includes pain items "Worst Pain in the Last Week", "Least Pain in the Last Week", and "Average Pain in the Last Week" and "Pain Right Now". Composite pain severity score (a mean severity score of the four pain items listed before). Composite pain interference score (a mean of the seven interference items). This will be calculated if at least four of the seven interference items have been completed on a given administration. Pain scores range from 0 to 10 with a score of 10 is the worst pain imaginable and a score of 0 is no pain. Worst observed scores is the highest score value observed.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 26
score on a scale
  Worst Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Worst Pain in the Last Week - Baseline | 4.0 (3.46)
  Least Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Least Pain in the Last Week - Baseline | 1.5 (1.81)
  Average Pain in the Last Week - Baseline: number analyzed (Participants) | 21
  Average Pain in the Last Week - Baseline | 2.4 (2.13)
  Pain Right Now - Baseline: number analyzed (Participants) | 21
  Pain Right Now - Baseline | 2.0 (1.99)
  Composite Pain Severity Score - Baseline: number analyzed (Participants) | 21
  Composite Pain Severity Score - Baseline | 2.476 (2.1779)
  Composite Pain Interference Score - Baseline: number analyzed (Participants) | 21
  Composite Pain Interference Score - Baseline | 2.869 (2.7136)
  Worst Pain in the Last Week - Overall Treatment Period | 6.7 (2.88)
  Least Pain in the Last Week - Overall Treatment Period | 3.9 (2.77)
  Average Pain in the Last Week - Overall Treatment Period | 4.9 (2.57)
  Pain Right Now - Overall Treatment Period | 5.1 (2.59)
  Composite Pain Severity Score - Overall Treatment Period | 4.885 (2.4374)
  Composite Pain Interference Score - Overall Treatment Period | 5.028 (2.9807)
  Worst Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Worst Pain in the Last Week - Change from Baseline in Overall Treatment Period | 2.4 (3.31)
  Least Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Least Pain in the Last Week - Change from Baseline in Overall Treatment Period | 2.0 (2.73)
  Average Pain in the Last Week - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Average Pain in the Last Week - Change from Baseline in Overall Treatment Period | 2.2 (2.59)
  Pain Right Now - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Pain Right Now - Change from Baseline in Overall Treatment Period | 2.9 (2.69)
  Composite Pain Severity Score - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Composite Pain Severity Score - Change from Baseline in Overall Treatment Period | 2.179 (2.6317)
  Composite Pain Interference Score - Change from Baseline in Overall Treatment Period: number analyzed (Participants) | 21
  Composite Pain Interference Score - Change from Baseline in Overall Treatment Period | 2.152 (2.9053)

5. Other Pre Specified Outcome: Number of Participants With Injection Site Reaction Adverse Events by Preferred Term
Description: Includes Adverse Events that have injection site reactions indicated as the Adverse Event High Level Terms
Time Frame: All AEs that are presented during or following initiation of trial treatment or worsens in severity are collected through the last scheduled visit (approximately 30 days after the last dose of treatment). Data were collected up to 29 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 29
Participants
  Injection site pain | 16
  Injection site erythema | 6
  Injection site induration | 4
  Injection site swelling | 4
  Injection site rash | 3
  Injection site discomfort | 2
  Injection site irritation | 1
  Injection site oedema | 1
  Injection site pruritus | 1

6. Other Pre Specified Outcome: Frequencies of Participants With Occurrence, Severity and Seriousness of Adverse Events
Description: Occurrence is defined as the number of participants who experienced an AE. Related SAEs are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per CTCAE v4.03 grade.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 29
Participants
  Treatment Emergent Adverse Events | 29
  Related Treatment Emergent Adverse Events | 28
  Severe Treatment Emergent Adverse Events | 11
  Severe Related Treatment Emergent Adverse Events | 3
  Serious Adverse Events | 8
  Related Serious Adverse Events | 2
  Adverse Events of Special Interest | 1
  Adverse Events Leading to Discontinuation | 1
  Adverse Events Leading to Death | 1
  Injection Site Reaction Adverse Events | 24

7. Other Pre Specified Outcome: Worst CTCAE Toxicity Grade Shift From Baseline in Laboratory Results (Hematology and Serum Chemistry)
Description: For hematology and chemistry laboratory parameters with CTCAE grading scales, toxicity grade shift is defined to evaluated categorical changes from baseline results to post-treatment results with respect to dichotomized CTCAE grading value (<= Grade 2, >= Grade 3). Grade 0=No adverse event or within normal limits; Grade 1=Mild adverse event; Grade 2=Moderate adverse event; Grade 3=Severe and undesirable adverse event; Grade 4=Life-threatening or disabling adverse event; Grade 5=Death related to adverse event. Higher scores mean worse outcome.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BN-Brachyury Plus Radiation
Number analyzed (Participants) | 29
Participants
  Hemoglobin: <= Grade 2 | 29
  Hemoglobin: >= Grade 3 | 0
  Hemoglobin: Missing | 0
  Leukocytes: <= Grade 2 | 29
  Leukocytes: >= Grade 3 | 0
  Leukocytes: Missing | 0
  Lymphocytes: <= Grade 2 | 23
  Lymphocytes: >= Grade 3 | 6
  Lymphocytes: Missing | 0
  Neutrophils: <= Grade 2 | 29
  Neutrophils: >= Grade 3 | 0
  Neutrophils: Missing | 0
  Platelets: <= Grade 2 | 29
  Platelets: >= Grade 3 | 0
  Platelets: Missing | 0
  Alanine Aminotransferase: <= Grade 2 | 29
  Alanine Aminotransferase: >= Grade 3 | 0
  Alanine Aminotransferase: Missing | 0
  Albumin: <= Grade 2 | 29
  Albumin: >= Grade 3 | 0
  Albumin: Missing | 0
  Alkaline Phosphatase: <= Grade 2 | 29
  Alkaline Phosphatase: >= Grade 3 | 0
  Alkaline Phosphatase: Missing | 0
  Aspartate Aminotransferase: <= Grade 2 | 29
  Aspartate Aminotransferase: >= Grade 3 | 0
  Aspartate Aminotransferase: Missing | 0
  Bilirubin: <= Grade 2 | 29
  Bilirubin: >= Grade 3 | 0
  Bilirubin: Missing | 0
  Calcium: <= Grade 2 | 29
  Calcium: >= Grade 3 | 0
  Calcium: Missing | 0
  Creatinine: <= Grade 2 | 29
  Creatinine: >= Grade 3 | 0
  Creatinine: Missing | 0
  Glucose: <= Grade 2 | 27
  Glucose: >= Grade 3 | 2
  Glucose: Missing | 0
  Magnesium: <= Grade 2 | 15
  Magnesium: >= Grade 3 | 0
  Magnesium: Missing | 14
  Phosphate: <= Grade 2 | 15
  Phosphate: >= Grade 3 | 0
  Phosphate: Missing | 14
  Potassium: <= Grade 2 | 29
  Potassium: >= Grade 3 | 0
  Potassium: Missing | 0
  Sodium: <= Grade 2 | 29
  Sodium: >= Grade 3 | 0
  Sodium: Missing | 0

ADVERSE EVENTS:
Time Frame: All Serious adverse events that are presented during or following initiation of trial treatment or worsens in severity after the initiation of trial treatment. They are collected through the last scheduled visit (approximately 30 days after the last dose of trial product). Data were collected up to 29 months.
Description: All Adverse events collected during or following initiation of trial treatment or worsens in severity after the initiation of trial treatment. They are collected through the last scheduled visit (approximately 30 days after the last dose of trial product). Data were collected up to 29 months.
Arm/Group | BN-Brachyury Plus Radiation
All-Cause Mortality (participants affected / at risk) | 2/29
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BN-Brachyury Plus Radiation (N=29)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BN-Brachyury Plus Radiation (N=29)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chills (General disorders) | 8 (10)
Fatigue (General disorders) | 16 (21)
Influenza like illness (General disorders) | 4 (5)
Injection site discomfort (General disorders) | 2 (2)
Injection site erythema (General disorders) | 6 (7)
Injection site induration (General disorders) | 4 (5)
Injection site pain (General disorders) | 16 (24)
Injection site rash (General disorders) | 3 (22)
Injection site swelling (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 3 (3)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 5 (7)
Urinary tract infection (Infections and infestations) | 5 (6)
Radiation skin injury (Injury, poisoning and procedural complications) | 8 (8)
Weight decreased (Investigations) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 7 (10)
Neuralgia (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03595228/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03595228/SAP_001.pdf